CLINICAL TRIAL: NCT00555126
Title: A Comparison of Forced-air With Endovascular Warming for Treatment of Accidental Hypothermia in Polytrauma Victims
Brief Title: Forced Air Versus Endovascular Warming in Polytrauma Patients
Acronym: FAEWPP
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Oliver Kimberger, Medical University of Vienna
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Polytrauma-007
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Polytrauma; Hypothermia
Keywords: Polytrauma; Hypothermia; Wound Infection; Blood Loss; Combined perioperative morbidity
MeSH Terms: conditions — Multiple Trauma; Hypothermia; Wound Infection; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warming with Forced Air (Active Comparator): Forced Air Warming
  Interventions: Device: Forced Air Warming
- Endovascular Warming (Experimental): Warming with Endovascular Catheter
  Interventions: Device: Warming with endovascular catheter + forced air warming

INTERVENTIONS:
Device: Forced Air Warming — Warming after Randomization
  Arms: Warming with Forced Air
Device: Warming with endovascular catheter + forced air warming — Warming after Randomization
  Arms: Endovascular Warming

SUMMARY:
Trauma is the leading cause of death in young adults, bleeding and infection are major concomitant problems. We test the hypothesis that fast, perioperative warming with an endovascular catheter versus forced air warming may improve patient outcome (primary outcome: combined perioperative morbidity, secondary outcome: bleeding, infection).

DETAILED DESCRIPTION:
Trauma is the leading cause of death in young adults and a major cause of morbidity and mortality at all ages. The acute problem is often uncontrollable bleeding. Subsequently, infection becomes a leading cause of morbidity. Polytrauma patients are at high risk for accidental hypothermia. Mild perioperative hypothermia causes a coagulopathy that significantly augments blood loss and increases allogeneic transfusion requirements. Hypothermia also impairs numerous immune functions - even slight decreases in core temperature triple the risk of surgical wound infection.

Endovascular temperature management system Alsius® (ICY, Alsius Corporation: Irvine,California,USA) has been approved in Europe and United States for the past 10 years and has been used in thousands of patients mainly for the indication of therapeutic cooling and subsequently rewarming of patients. A major potential advantage of this system is that heat is directly added to the thermal core, thus bypassing the heat sink and insulating effects of peripheral tissues. The efficacy of this system is sufficient to allow rapid rewarming in hypothermic trauma victims, even those undergoing major surgery. We therefore propose to test the hypothesis that polytrauma patients rewarmed with the Alsius® system will have better patient outcome (combined perioperative morbidity) than those warmed conventionally with forced-air.

ELIGIBILITY:
Inclusion Criteria:

We will evaluate patients admitted to the Emergency department for polytrauma. Patients will be eligible for the study when they:

1. Are between 18 and 70 years old
2. Have a Glasgow coma score ≥ 9
3. An ISS (Injury Severity Score) ≥16; and
4. Have A Severity Characterisation Of Trauma (ASCOT) score predicting mortality ranging from 2 to 50% (www.sfar.org/scores2/ascot2.html).

Exclusion Criteria:

Patients will be excluded if they are:

1. <150cm in height
2. Known to have a vena cava filter
3. Known to have a history of coagulopathy including anti-coagulant medications; or
4. Known to be pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Combined Perioperative Morbidity | During LOS (approximately 30 days)

SECONDARY OUTCOMES:
Blood Loss | Perioperative Period
Infection | Perioperative Period, during LOS

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, M.D., Principal Investigator — Medical University of Vienna
Locations (2):
- Austria (2):
  - Medical University of Vienna, Vienna, Vienna
  - Lorenz Böhler Unfallkrankenhaus, Vienna, Vienna

REFERENCES:
- [Background] Greif R, Akca O, Horn EP, Kurz A, Sessler DI; Outcomes Research Group. Supplemental perioperative oxygen to reduce the incidence of surgical-wound infection. N Engl J Med. 2000 Jan 20;342(3):161-7. doi: 10.1056/NEJM200001203420303. PMID 10639541
- [Background] Winkler M, Akca O, Birkenberg B, Hetz H, Scheck T, Arkilic CF, Kabon B, Marker E, Grubl A, Czepan R, Greher M, Goll V, Gottsauner-Wolf F, Kurz A, Sessler DI. Aggressive warming reduces blood loss during hip arthroplasty. Anesth Analg. 2000 Oct;91(4):978-84. doi: 10.1097/00000539-200010000-00039. PMID 11004060